CLINICAL TRIAL: NCT05838560
Title: Dasatinib Plus Quercetin for Accelerated Aging in Mental Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: UConn Health (Other)
Responsible Party: Principal Investigator, Eric Lenze, Wallace and Lucille K Renard Prof of Psychiatry, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202302203
Record Dates: First submitted 2023-04-17; First posted 2023-05-01 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia; Treatment Resistant Depression; Aging, Premature
Keywords: Schizophrenia; Treatment Resistant Depression; Aging, Premature; Older Adults
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Treatment-Resistant; Aging, Premature | interventions — Dasatinib; Quercetin

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dasatinib + quercetin (Experimental): open label dasatinib plus quercetin combined as a drug therapy
  Interventions: Drug: Dasatinib; Drug: quercetin

INTERVENTIONS:
Drug: Dasatinib — dasatinib 100mg The intervention will involve the participant taking dasatinib 100mg and quercetin 1250ng combined.
  Other Names: sprycel; sophoretin
Drug: quercetin — The intervention will involve the participant taking dasatinib 100mg and quercetin 1250ng combined.
  Other Names: quercetine; Vitamine P

SUMMARY:
This pilot open-label study examines the effects of a combination of dasatinib plus quercetin - two drugs that have known senolytics properties - on physiological aging in older individuals with depression or schizophrenia.

DETAILED DESCRIPTION:
This is a pilot study that will enroll up to 40 participants and will examine the following:

1. test the safety and feasibility of dasatinib+quercetin in two mental illnesses associated with accelerated aging: schizophrenia and treatment-resistant depression
2. examine changes in SASP (senescence-associated secretory phenotype) with dasatinib+quercetin treatment
3. examine acute and long-term changes in neuropsychological functioning, functional status, and brain markers of aging, as well as in clinical symptoms of the illnesses (treatment-resistant depression and schizophrenia).

This study will also combine the treatment of dasatinib plus quercetin and lifestyle-based risk factor management - which will involve the research team during the medication intervention portion to provide lifestyle education focusing on strength, balance, and nutrition. The research team will maintain close contact with participants to offer encouragement, address questions and help navigate barriers to engaging in the activities.

Before study enrollment, participants will be screened using questionnaires and a phone screen prior to being consented.

The participant will be involved for about 1 year and self-administer 8 total doses of the medications - two consecutive days of dasatinib 100mg orally plus quercetin 1250mg orally on weeks 1 (ie., 2 days on, 5 days off), 2, 3, and 4.

The participant will undergo an MRI scan at baseline and approximately week 10 of the study.

Blood draws will occur at baseline, week 1, 2, 3, 4, 10, and at the endpoint. 10 ml of blood will be taken each time for 700 ml over 1 year.

Participants will have several questionnaires and assessments to complete at baseline, week 10, and the study's endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Either major depression, which is treatment-resistant (currently depressed despite at least 2 adequate trials of antidepressants in this or the previous episode), or schizophrenia/schizoaffective disorder.
2. Age 50+ (60+ for depression).
3. Three conditions associated with aging (e.g., hypertension/diabetes/metabolic syndrome, cardiac disease, lung disease other than asthma, cancer with adult-onset, arthritis, and inflammatory diseases typically seen in aging).
4. No history of dementia by patient report.
5. Already taking an adequate dose of medication for schizophrenia/schizoaffective disorder or depression.

Exclusion Criteria:

1. Contraindications for dasatinib or quercetin
2. Active SI such that participant could not be safely managed in an outpatient clinical trial.
3. Taking medications that are strong CPY3A4 inhibitors or strong inducers, or that induce senescence (e.g., alkylating agents, anthracyclines, platins/other chemotherapy), or everolimus and topotecan (which have interactions with quercetin).
4. All medications and medical conditions will be reviewed by physician study investigators to determine whether the medication or condition, in the opinion of the investigators, makes the participant inappropriate for the study. Examples of such potential excluding conditions: Active inflammatory, infectious, or malignant disease; sensory deficits that would interfere with assessments; recent heart attack or stroke; severe bleeding disorder; uncontrolled hypertension or diabetes mellitus; active liver disease or cirrhosis; current use of systemic steroids, quinolone antibiotics, hydroxychloroquine or chloroquine.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who successfully completed and safely tolerated the intervention | 10 weeks
  Test the safety and feasibility of dasatinib plus quercetin

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lenze, MD, Principal Investigator — Washington University School of Medicine, Department of Psychiatry
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data available upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available by request within 1 year of the final data collection.
Access Criteria: Contact study PI

REFERENCES:
- [Derived] Schweiger A, Diniz B, Nicol G, Schweiger J, Dasklakis-Perez AE, Lenze EJ. Protocol for a pilot clinical trial of the senolytic drug combination Dasatinib Plus Quercetin to mitigate age-related health and cognitive decline in mental disorders. F1000Res. 2025 Mar 5;13:1072. doi: 10.12688/f1000research.151963.2. eCollection 2024. PMID 40443429